CLINICAL TRIAL: NCT02176980
Title: Hepatitis C Alcohol Reduction Treatment - Randomized Controlled Trial (Hep ART-RCT)
Brief Title: Hepatitis C Alcohol Reduction Treatment
Acronym: HepART-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00046518
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C, Chronic; AUD
Keywords: HCV; hepatitis C; alcohol; integrated care
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — Ethanol; Counseling; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical provider (MP) brief alcohol counseling & referral (Active Comparator): 1. Screening of HCV-infected patients for alcohol use using the 10-item Alcohol Use Disorders Identification Test (AUDIT).
  2. Patients self-administer the AUDIT.
  3. HCV providers review the AUDIT with the patient.
  4. If the patient is using any alcohol, the HCV provider conducts brief alcohol counseling using the FRAMES model, based on the evidence-based Screening, Brief Intervention, and Referral to Treatment (SBIRT) method.
  5. Medical provider will explain the importance of alcohol abstinence in the presence of HCV infection.
  6. Patient is referred to an alcohol treatment programs outside the liver clinic. Typical counseling will take the form of individual and group therapy.
  Interventions: Behavioral: Brief alcohol counseling
- Brief alcohol counseling & 6 months of HCV-alcohol treatment (Experimental): * Steps 1 through 5 as described in comparator arm above.
  * 6 months of group therapy, offered weekly.
  * 6 months of individual therapy, in person or by phone, offered every two weeks.
  * Therapy content emphasizes interplay between alcohol use and liver health/HCV.
  * Informal collaboration between HCV providers and addictions therapists.
  * Shared EMR charting.
  * Referral to study-provided psychiatry as needed.
  Interventions: Behavioral: Group and Individual Therapy Sessions

INTERVENTIONS:
Behavioral: Brief alcohol counseling — Medical provider gives feedback on how the patient's alcohol use may affect their current and future health, noting that it is the patient's responsibility to change behavior; giving advice to stop drinking based on medical concern; giving a menu of options for cutting down on drinking; expressing empathy; and reinforcing the patient's self-efficacy to change.
  Arms: Medical provider (MP) brief alcohol counseling & referral
Behavioral: Group and Individual Therapy Sessions — Session content integrates HCV and alcohol issues in treatment, liver health, and personal realms. Sessions include psychoeducational content on how alcohol affects the liver among people with HCV; HCV stigma; family issues around drinking and the HCV diagnosis; nutrition; life goals and positive affect; and alcohol reduction strategies.
  Arms: Brief alcohol counseling & 6 months of HCV-alcohol treatment

SUMMARY:
Subjects are being asked to take part in a research study to test two levels of alcohol services for patients with hepatitis C virus (HCV) who drink alcohol. The two levels differ in intensity of alcohol services and in whether or not they include a focus on liver health. The study will look at which level of alcohol services best decreases alcohol use among patients with HCV.

DETAILED DESCRIPTION:
For people infected with hepatitis C virus (HCV), alcohol use increases the risk of hepatocellular carcinoma and progressive liver fibrosis, which can lead to cirrhosis and liver-related mortality. Integrated models of care that incorporate treatment for alcohol use, substance use, and mental health comorbidities have been called for, but few empirically tested models exist.

In an R21 study, we developed and manualized an integrated behavioral-medical treatment model for patients with HCV who consume alcohol. Investigators successfully implemented a standardized alcohol screening in a liver clinic using the Alcohol Use Disorders Identification Test (AUDIT) instrument; recruited 60 patients; retained participants in group and individual therapy; integrated care between an addictions therapist and medical providers; and achieved an 85% six-month interview response rate. The alcohol abstinence rate improved from 0% at baseline to 44% at 6 months. Mean Addiction Severity Index scores were reduced by 50% for alcohol from .24 to .12, and decreased for drug use from .05 to .03. The percentage of heavy drinkers decreased from 47% to 24% (Proeschold-Bell et al., 2011).

This study will conduct a randomized controlled trial that compares medical provider-delivered brief alcohol counseling plus our on-site six-month integrated treatment to brief alcohol counseling plus outside alcohol treatment referral in 279 HCV-infected patients with qualifying AUDIT alcohol scores at baseline. Participants in both arms will be treated at the Duke and UNC Liver Clinics and the Durham Veterans Affairs Medical Center. Outcome variables will be assessed at baseline, 3, 6, and 12 months. The aims are to 1) evaluate alcohol abstinence; 2) determine differences in secondary outcomes between study arms; and 3) conduct a cost effectiveness analysis. Investigators hypothesize that the intervention will significantly improve alcohol abstinence rates and significantly decrease relapse rates compared to the comparison. Investigators further hypothesize that intervention participants will report fewer drinks per week than comparison participants, have fewer positive drug screens than comparison participants, and meet the $50,000 per quality-adjusted life year gained standard established in the health economics literature.

ELIGIBILITY:
Inclusion criteria

* Ever HCV-infected chronic HCV
* Appropriate score on the Alcohol Use Disorder Identification Test (AUDIT)

  * Females, ≥4
  * Males, ≥8
* Consumed alcohol in past 60 days
* Not currently attending alcohol treatment services more than once every two weeks. If you attend treatment services at least once every two weeks, you must have either drunk alcohol heavily in the past 2 weeks or have drunk alcohol at least 7 of the past 14 days or your medical provider must have assessed that you would benefit from alcohol treatment services offered by this study

  * Patient at one of the 3 clinic sites
* 18 or older
* English-speaking
* OK to have HIV, substance use or other co-morbidities, or receiving HCV antiviral treatment

Exclusion criteria

* Psychotic
* Insurmountable transportation barriers (can receive individual therapy by phone but need appointments with HCV provider at 3 and 6 months and ideally some in-person group therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-10; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Alcohol abstinence rates at 6 months after consent | 6 months
  Investigators will compare the two treatment arms on occurrence and amount of past 180 days of drinking using the timeline follow-back method, allowing the investigators to assess change in number of drinking days, periods of abstinence, and total grams of alcohol consumed.

SECONDARY OUTCOMES:
Relapse rate at 12 months after consent | 12 months
  Investigators will compare the two treatment arms on periods of abstinence and number of drinking days using the timeline follow-back method for the 180 days between 6 and 12 months since study consent.
Other alcohol use indicators | 3, 6 and 12 months
  At 3, 6 and 12 months, investigators will assess the number of heavy drinking days and grams of alcohol consumed and compare between the two treatment arms.
Illicit drug use | 3, 6 and 12 months
  At 3, 6 and 12 months, investigators will assess illicit drug use based on positive/negative urine toxicology screens and compare between the two treatment arms.

OTHER OUTCOMES:
Cost effectiveness analysis of the intervention versus brief alcohol counseling and referral out | 12 months
  The incremental cost-effectiveness ratio (ICER) will be absolute difference in costs divided by the absolute difference in various effectiveness measures between the 2 interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Muir, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Proeschold-Bell RJ, Patkar AA, Naggie S, Coward L, Mannelli P, Yao J, Bixby P, Muir AJ. An integrated alcohol abuse and medical treatment model for patients with hepatitis C. Dig Dis Sci. 2012 Apr;57(4):1083-91. doi: 10.1007/s10620-011-1976-4. Epub 2011 Dec 2. PMID 22134784
- [Background] Proeschold-Bell RJ, Evon DM, Makarushka C, Wong JB, Datta SK, Yao J, Patkar AA, Mannelli P, Hodge T, Naggie S, Wilder JM, Fried MW, Niedzwiecki D, Muir AJ. The Hepatitis C-Alcohol Reduction Treatment (Hep ART) intervention: Study protocol of a multi-center randomized controlled trial. Contemp Clin Trials. 2018 Sep;72:73-85. doi: 10.1016/j.cct.2018.07.003. Epub 2018 Jul 10. PMID 30006024